CLINICAL TRIAL: NCT03399045
Title: Impact of 9-minute Withdrawal Time on Adenoma Detection Rate：a Multicenter, Prospective, Randomized Controlled Trial
Brief Title: 9 Minutes for Colonoscopy Withdrawal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Changhai Hospital (Other)
Collaborators: No.85 Hospital, Changning, Shanghai, China (Other); The Second Clinical Medical College of Jinan University (Other); Qinghai People's Hospital (Other); Shaanxi Provincial People's Hospital (Other); Shanghai 8th People's Hospital (Other); Yantaishan Hospital of Yantai City (Unknown); First Affiliated Hospital of Harbin Medical University (Other); Changzhi People's Hospital (Other); Ningbo Medical Center Li Huili Eastern Hospital (Unknown); The Third People's Hospital of Datong (Unknown); The First Affiliated Hospital of the Medical College, Shihezi University (Unknown); The First Affiliated Hospital of Dalian Medical University (Other); Seventh Medical Center of PLA Army General Hospital (Other)
Responsible Party: Principal Investigator, Zhaoshen Li, Director of Gastroenterology Dept, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: withdrawal time-1
Record Dates: First submitted 2018-01-08; First posted 2018-01-16 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Colon Polyps; Colorectal Adenomas
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 9-minute withdrawal group (Experimental): Patients in 9-minute withdrawal group will be carefully observed for 9 minutes during the colonoscopy withdraw. A stop watch will be utilized to remind endoscopists the withdrawal time. The time to perform polyp biopsy will not be included in the 9 minutes.
  Interventions: Procedure: 9-minute withdrawal
- 6-minute withdrawal group (Active Comparator): Patients in 6-minute withdrawal group will be carefully observed for 6 minutes during the colonoscopy withdraw. A stop watch will be utilized to remind endoscopists the withdrawal time. The time to perform polyp biopsy willwill not be included in the 9 minutes.
  Interventions: Procedure: 6-minute withdrawal

INTERVENTIONS:
Procedure: 9-minute withdrawal — Patients in 9-minute withdrawal group will be carefully observed for 9 minutes during the colonoscopy withdraw
  Arms: 9-minute withdrawal group
Procedure: 6-minute withdrawal — Patients in 6-minute withdrawal group will be carefully observed for 6 minutes during the colonoscopy withdraw
  Arms: 6-minute withdrawal group

SUMMARY:
A withdrawal time of at least 6 minutes has been considered to be necessary to guarantee the adenoma detection rate and the critical quality criterion of colonoscopy. However, several large observational investigations demonstrated that 9 minutes will be in favor of higher adenoma detection rate and lower risk of interval colorectal cancer, when compared with 6-minute withdrawal. Meanwhile, a few studies also indicated that no significant benefit were observed in longer withdrawal time. Up to now, no randomized controlled trials have been conducted to give a definitive conclusion. Therefore, we performed a multicenter, prospective, randomized Controlled trial to compare adenoma detection rate of 6-minute and 9-minute withdrawal in colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Patients whose age is between 40-85.
* Patients who have indications for screening, surveillance and diagnostic colonoscopy.
* Patients who have signed inform consent form

Exclusion Criteria:

* Patients who have undergone colonic resection
* Patients with intracranial and/or central nervous system disease, including cerebral infarction and cerebral hemorrhage.
* Patients with severe chronic cardiopulmonary and renal disease.
* Patients who are unwilling or unable to consent.
* Patients who are not suitable for colonoscopy
* Patients who received urgent or therapeutic colonoscopy
* Patients with pregnancy, inflammatory bowel disease, polyposis of colon, colorectal cancer, or intestinal obstruction
* Patients who are taking aspirin, clopidogrel or other anticoagulants
* Patients with Aronchick score > 3

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1027 (Actual)
Dates: Start 2018-01-20 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-06 (Actual)

PRIMARY OUTCOMES:
adenoma detection rate(ADR) | 30mins
  ADR was calculated adenoma detection rate is the number of patients with at least one adenoma, divided by the total number of patients.

SECONDARY OUTCOMES:
adenomas per colonoscopy(APC) | 30mins
  APC was calculated as the number of adenomas detected during colonoscopy withdraw divided by the number of colonoscopies.

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhaoshen, M.D, Principal Investigator — Changhai Hospital
Locations (1):
- Changhai Hospital, Second Military Medical University, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zhao S, Yang X, Wang S, Meng Q, Wang R, Bo L, Chang X, Pan P, Xia T, Yang F, Yao J, Zheng J, Sheng J, Zhao X, Tang S, Wang Y, Wang Y, Gong A, Chen W, Shen J, Zhu X, Wang S, Yan C, Yang Y, Zhu Y, Ma RJ, Wang R, Ma Y, Li Z, Bai Y. Impact of 9-Minute Withdrawal Time on the Adenoma Detection Rate: A Multicenter Randomized Controlled Trial. Clin Gastroenterol Hepatol. 2022 Feb;20(2):e168-e181. doi: 10.1016/j.cgh.2020.11.019. Epub 2020 Nov 19. PMID 33220526